CLINICAL TRIAL: NCT03656718
Title: Phase I/II Pharmacokinetic Multi-Tumor Study of Subcutaneous Formulation of Nivolumab Monotherapy
Brief Title: A Study of Subcutaneous Nivolumab Monotherapy With or Without Recombinant Human Hyaluronidase PH20 (rHuPH20)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA209-8KX; 2018-001585-42 (EudraCT Number)
Record Dates: First submitted 2018-08-28; First posted 2018-09-04 (Actual); Results first posted 2025-02-20 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-10

CONDITIONS: Neoplasms by Site
Keywords: Subcutaneous; Nivolumab; rHuPH20
MeSH Terms: conditions — Neoplasms by Site | interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Part A, Group 1: nivolumab (dose 1) + rHuPH20 (Experimental)
  Interventions: Biological: nivolumab; Drug: rHuPH20
- Part B, Group 3: nivolumab (dose 2) + rHuPH20 (Experimental)
  Interventions: Biological: nivolumab; Drug: rHuPH20
- Part B, Group 2: nivolumab (dose 1) (Experimental)
  Interventions: Biological: nivolumab
- Part B, Group 4: nivolumab (dose 2) (Experimental)
  Interventions: Biological: nivolumab
- Part C: nivolumab (dose 3) + rHuPH20 (Experimental)
  Interventions: Biological: nivolumab; Drug: rHuPH20
- Part D, Group 5: nivolumab (dose 3) + rHuPH20 (Experimental)
  Interventions: Biological: nivolumab; Drug: rHuPH20
- Part E, Group 6: nivolumab (dose 4) coformulated with rHuPH20 (Experimental)
  Interventions: Biological: nivolumab; Drug: rHuPH20

INTERVENTIONS:
Biological: nivolumab — (Subcutaneous) Specified dose on specified days
  Other Names: Opdivo; BMS-986298
Drug: rHuPH20 — Specified dose on specified days Permeation enhancer
  Other Names: ENHANZE™ DP
  Arms: Part A, Group 1: nivolumab (dose 1) + rHuPH20; Part B, Group 3: nivolumab (dose 2) + rHuPH20; Part C: nivolumab (dose 3) + rHuPH20; Part D, Group 5: nivolumab (dose 3) + rHuPH20; Part E, Group 6: nivolumab (dose 4) coformulated with rHuPH20
Biological: nivolumab — (IV) Specified Dose on Specified Days
  Other Names: BMS-936558
  Arms: Part A, Group 1: nivolumab (dose 1) + rHuPH20; Part B, Group 2: nivolumab (dose 1); Part B, Group 3: nivolumab (dose 2) + rHuPH20; Part B, Group 4: nivolumab (dose 2)

SUMMARY:
The purpose of this study is to investigate the effects of nivolumab when given under the skin with or without rHuPH20.

This study will include participants with 1 of the following advanced or metastatic tumors approved for treatment with nivolumab monotherapy:

* non-small cell lung cancer (NSCLC)
* renal cell carcinoma (RCC)
* unresectable or metastatic melanoma
* hepatocellular carcinoma (HCC)
* microsatellite instability-high or mismatch repair deficient colorectal cancer (MSI-H/dMMR CRC)
* in Part B, other solid tumors may be considered at the discretion of the Clinical Trial Physician
* In addition to the above tumors, Part E will also include participants with metastatic urothelial carcinoma (mUC).

ELIGIBILITY:
Inclusion Criteria:

* Histologic or cytologic confirmation of advanced (metastatic and/or unresectable) solid tumors of one of the following tumor types:

  1. Metastatic squamous or non-squamous NSCLC
  2. RCC, advanced or metastatic
  3. Melanoma
  4. HCC
  5. CRC, metastatic (MSI-H or dMMR)
  6. In Part B, other solid tumor types may be considered at the discretion of the Medical Monitor
  7. In Part E, Metastatic urothelial carcinoma
* Measurable disease as per RECIST version 1.1 criteria
* ECOG performance status of 0 or 1

Exclusion Criteria:

* Active brain metastases or leptomeningeal metastases
* Ocular melanoma
* Active, known, or suspected autoimmune disease

Other protocol defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2018-10-29 (Actual); Primary Completion 2022-09-07 (Actual); Study Completion 2024-09-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (36):
- United States (10):
  - Winship Cancer Institute., Atlanta, Georgia
  - Local Institution - 0024, Rockville, Maryland
  - Local Institution - 0020, Detroit, Michigan
  - Local Institution - 0001, Charlotte, North Carolina
  - Local Institution - 0012, Eugene, Oregon
  - Greenville Health System, Greenville, South Carolina
  - Local Institution - 0010, Austin, Texas
  - Local Institution - 0009, Beaumont, Texas
  - Local Institution - 0007, Dallas, Texas
  - Local Institution - 0011, Tyler, Texas
- Argentina (2):
  - Local Institution - 0035, CABA
  - Local Institution - 0025, CABA
- Brazil (2):
  - Local Institution - 0038, Porto Alegre, Rio Grande do Sul
  - Local Institution - 0037, São Paulo
- Local Institution - 0005, Santiago, Chile
- France (2):
  - Local Institution - 0022, Saint-Herblain
  - Local Institution - 0021, Villejuif
- Italy (2):
  - Local Institution - 0003, Rozzano, MI
  - Local Institution - 0004, Padua
- Mexico (6):
  - Local Institution - 0050, Mexico City, Mexico City
  - Local Institution - 0048, Mexico City, Mexico City
  - Local Institution - 0046, Monterrey, Nuevo León
  - Local Institution - 0047, Monterrey, Nuevo León
  - Local Institution - 0049, Puebla City
  - Local Institution - 0045, Querétaro
- Netherlands (2):
  - Local Institution - 0026, Amsterdam, North Holland
  - Local Institution - 0039, Maastricht
- New Zealand (4):
  - Local Institution - 0040, Rotorua, Bay of Plenty
  - Local Institution - 0018, Newtown, Wellington Region
  - Local Institution - 0014, Dunedin
  - Local Institution - 0015, Tauranga
- Local Institution - 0019, Warsaw, Masovian Voivodeship, Poland
- Spain (2):
  - Local Institution - 0017, Madrid
  - Local Institution - 0016, Málaga
- United Kingdom (2):
  - Local Institution - 0033, Cardiff, Glamorgan
  - Local Institution - 0031, Liverpool

REFERENCES:
- [Derived] Lonardi S, Lugowska I, O'Donnell A, Jackson C, Latten-Jansen LM, North R, Bahleda R, Garrido M, Santoro A, Chacon MR, Li L, Joseph D, Vezina HE, Aras U, Bennett B, Perumal D, Gurm B, Ng WT, Harvey RD, Trigo J, Calvo A. Pharmacokinetics and safety of subcutaneous nivolumab: results from the phase I/II CheckMate 8KX study. J Immunother Cancer. 2025 Oct 5;13(10):e011918. doi: 10.1136/jitc-2025-011918. PMID 41052885
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.BMSClinicalTrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 28 participants from Part A and Part B crossed over after completing treatment in their originally assigned Arms to form Part C.
Groups:
- Part A - Group 1: Nivolumab + rHuPH20 SC 720mg: Single dose of nivolumab (BMS-986298) 720 mg administered subcutaneously (SC) with recombinant human hyaluronidase (rHuPH20) manually by syringe. Four weeks after the single nivolumab SC (BMS-986298) dose participants received IV nivolumab (BMS-936558) 480 mg Q4W dosing until Response Evaluation Criteria in Solid Tumors (RECIST) v.1.1 progression, unacceptable toxicity, withdrawal of consent, completion of 104 weeks of treatment, cross over to nivolumab SC dosing in Part C whichever occurred first. In certain circumstances, participants with progressive disease per RECIST v1.1 but with otherwise stable or improved performance and clinical status could continue to be treated in the event of a perceived benefit per Investigator.
- Part B - Group 2: Nivolumab SC 720mg: Single dose of nivolumab (BMS-986298) 720 mg administered subcutaneously (SC) without recombinant human hyaluronidase (rHuPH20) by syringe pump. Four weeks after the single nivolumab SC (BMS-986298) dose participants received IV nivolumab (BMS-936558) 480 mg Q4W dosing until Response Evaluation Criteria in Solid Tumors (RECIST) v.1.1 progression, unacceptable toxicity, withdrawal of consent, completion of 104 weeks of treatment, cross over to nivolumab SC dosing in Part C, whichever occurred first. In certain circumstances, participants with progressive disease per RECIST v1.1 but with otherwise stable or improved performance and clinical status could continue to be treated in the event of a perceived benefit per Investigator.
- Part B - Group 3: Nivolumab + rHuPH20 SC 960mg: Single dose of nivolumab (BMS-986298) 960 mg administered subcutaneously (SC) with recombinant human hyaluronidase (rHuPH20) manually by syringe. Four weeks after the single nivolumab SC (BMS-986298) dose participants received IV nivolumab (BMS-936558) 480 mg Q4W dosing until Response Evaluation Criteria in Solid Tumors (RECIST) v.1.1 progression, unacceptable toxicity, withdrawal of consent, completion of 104 weeks of treatment, cross over to nivolumab SC dosing in Part C, whichever occurred first. In certain circumstances, participants with progressive disease per RECIST v1.1 but with otherwise stable or improved performance and clinical status could continue to be treated in the event of a perceived benefit per Investigator.
- Part B - Group 4: Nivolumab SC 960mg: Single dose of nivolumab (BMS-986298) 960 mg administered subcutaneously (SC) without recombinant human hyaluronidase (rHuPH20) by syringe pump. Four weeks after the single nivolumab SC (BMS-986298) dose participants received IV nivolumab (BMS-936558) 480 mg Q4W dosing until Response Evaluation Criteria in Solid Tumors (RECIST) v.1.1 progression, unacceptable toxicity, withdrawal of consent, completion of 104 weeks of treatment, cross over to nivolumab SC dosing in Part C, whichever occurred first. In certain circumstances, participants with progressive disease per RECIST v1.1 but with otherwise stable or improved performance and clinical status could continue to be treated in the event of a perceived benefit per Investigator.
- Part C - Nivolumab SC + rHuPH20 1200 mg Q4W: Some participants in Part A and Part B crossed over to Part C, four weeks after their last nivolumab IV dose to receive nivolumab (BMS-986298) 1200 mg administered subcutaneously (SC) with recombinant human hyaluronidase (rHuPH20) manually by syringe every 4 weeks. Treatment continued until Response Evaluation Criteria in Solid Tumors (RECIST) v.1.1 progression, unacceptable toxicity, withdrawal of consent, or completion of 104 weeks of treatment, whichever occurred first. In certain circumstances, participants with progressive disease per RECIST v1.1 but with otherwise stable or improved performance and clinical status could continue to be treated in the event of a perceived benefit per Investigator.
- Part D: Nivolumab SC + rHuPH20 SC 1200mg Q4W: Nivolumab (BMS-986298) 1200 mg administered subcutaneously (SC) with recombinant human hyaluronidase (rHuPH20) manually by syringe every 4 weeks. Treatment continued until Response Evaluation Criteria in Solid Tumors (RECIST) v.1.1 progression, unacceptable toxicity, withdrawal of consent, or completion of 104 weeks of treatment, whichever occurred first. In certain circumstances, participants with progressive disease per RECIST v1.1 but with otherwise stable or improved performance and clinical status could continue to be treated in the event of a perceived benefit per Investigator.
- Part E: Nivolumab SC Co-Formulated With rHuPH20 600mg Q2W: Nivolumab (BMS-986298) 600 mg coformulated with recombinant human hyaluronidase (rHuPH20) administered subcutaneously (SC) manually by syringe every 2 weeks. Treatment continued until Response Evaluation Criteria in Solid Tumors (RECIST) v.1.1 progression, unacceptable toxicity, withdrawal of consent, or completion of 104 weeks of treatment, whichever occurred first. In certain circumstances, participants with progressive disease per RECIST v1.1 but with otherwise stable or improved performance and clinical status could continue to be treated in the event of a perceived benefit per Investigator.
Period: Pre-Treatment Period
Arm/Group | Part A - Group 1: Nivolumab + rHuPH20 SC 720mg | Part B - Group 2: Nivolumab SC 720mg | Part B - Group 3: Nivolumab + rHuPH20 SC 960mg | Part B - Group 4: Nivolumab SC 960mg | Part C - Nivolumab SC + rHuPH20 1200 mg Q4W | Part D: Nivolumab SC + rHuPH20 SC 1200mg Q4W | Part E: Nivolumab SC Co-Formulated With rHuPH20 600mg Q2W
Started | 22 | 18 | 10 | 17 | 0 | 36 | 36
Completed | 22 | 18 | 10 | 17 | 0 | 36 | 36
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Treatment Period Parts A, B, D, and E
Arm/Group | Part A - Group 1: Nivolumab + rHuPH20 SC 720mg | Part B - Group 2: Nivolumab SC 720mg | Part B - Group 3: Nivolumab + rHuPH20 SC 960mg | Part B - Group 4: Nivolumab SC 960mg | Part C - Nivolumab SC + rHuPH20 1200 mg Q4W | Part D: Nivolumab SC + rHuPH20 SC 1200mg Q4W | Part E: Nivolumab SC Co-Formulated With rHuPH20 600mg Q2W
Started | 22 | 18 | 10 | 17 | 0 | 36 | 36
Completed | 10 | 6 | 5 | 9 | 0 | 7 | 6
Not Completed | 12 | 12 | 5 | 8 | 0 | 29 | 30
Not completed — Disease progression | 8 | 11 | 4 | 6 | 0 | 20 | 21
Not completed — Study drug toxicity | 2 | 1 | 1 | 2 | 0 | 4 | 1
Not completed — Death | 1 | 0 | 0 | 0 | 0 | 0 | 2
Not completed — Adverse event unrelated to study drug | 0 | 0 | 0 | 0 | 0 | 4 | 1
Not completed — Participant requested to discontinue study treatment | 1 | 0 | 0 | 0 | 0 | 0 | 2
Not completed — Other reasons | 0 | 0 | 0 | 0 | 0 | 1 | 3
Period: Treatment Period Part C
Arm/Group | Part A - Group 1: Nivolumab + rHuPH20 SC 720mg | Part B - Group 2: Nivolumab SC 720mg | Part B - Group 3: Nivolumab + rHuPH20 SC 960mg | Part B - Group 4: Nivolumab SC 960mg | Part C - Nivolumab SC + rHuPH20 1200 mg Q4W | Part D: Nivolumab SC + rHuPH20 SC 1200mg Q4W | Part E: Nivolumab SC Co-Formulated With rHuPH20 600mg Q2W
Started | 0 | 0 | 0 | 0 | 28 (9 Participants crossed over from Part A - Group 1, 6 participants crossed over from Part B -Group 2, 5 participants crossed over from Part B -Group 3, 8 participants crossed over from Part B -Group 4.) | 0 | 0
Completed | 0 | 0 | 0 | 0 | 12 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 16 | 0 | 0
Not completed — Disease progression | 0 | 0 | 0 | 0 | 12 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Participant requested to discontinue study treatment | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Other reasons | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Maximum clinical benefit | 0 | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Participants in Part C are presented under their original treatment assignment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A - Group 1: Nivolumab + rHuPH20 SC 720mg | Part B - Group 2: Nivolumab SC 720mg | Part B - Group 3: Nivolumab + rHuPH20 SC 960mg | Part B - Group 4: Nivolumab SC 960mg | Part D: Nivolumab SC + rHuPH20 SC 1200mg Q4W | Part E: Nivolumab SC Co-Formulated With rHuPH20 600mg Q2W | Total
Number analyzed (Participants) | 22 | 18 | 10 | 17 | 36 | 36 | 139
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 12 | 5 | 6 | 14 | 19 | 62
  >=65 years | 16 | 6 | 5 | 11 | 22 | 17 | 77
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 5 | 6 | 5 | 10 | 9 | 47
  Male | 10 | 13 | 4 | 12 | 26 | 27 | 92
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 0 | 4 | 1 | 6
  Not Hispanic or Latino | 4 | 5 | 2 | 7 | 16 | 22 | 56
  Unknown or Not Reported | 17 | 13 | 8 | 10 | 16 | 13 | 77
Race/Ethnicity, Customized [Number; unit: Participants] — Race
  Participants
    White | 18 | 18 | 8 | 17 | 31 | 34 | 126
    Black or African American | 2 | 0 | 0 | 0 | 1 | 0 | 3
    Other | 2 | 0 | 2 | 0 | 3 | 1 | 8
    Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Asian | 0 | 0 | 0 | 0 | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Serum Nivolumab Concentration (Cmax) - Parts A, B, D, and E
Description: Cmax is the maximum observed serum nivolumab concentration. Collected for Arm A, B, and D on Cycle 1 Day 1, Cycle 1 Day 2, Cycle 1 Day 4, Cycle 1 Day 8, Cycle 1 Day 15, and Cycle 1 Day 21. Collected for Arm E on Cycle 1 Day 1, Cycle 1 Day 2, Cycle 1 Day 4, Cycle 1 Day 8, Cycle 1 Day 15.
Time Frame: From first dose until approximately 21 days post first dose.
Population: All treated participants with available Cycle 1 PK results in Parts A, B, D, and E. Pre-specified for data to be reported for Parts A, B, D, and E only.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Part A - Group 1: Nivolumab + rHuPH20 SC 720mg | Part B - Group 2: Nivolumab SC 720mg | Part B - Group 3: Nivolumab + rHuPH20 SC 960mg | Part B - Group 4: Nivolumab SC 960mg | Part D: Nivolumab SC + rHuPH20 SC 1200mg Q4W | Part E: Nivolumab SC Co-Formulated With rHuPH20 600mg Q2W
Number analyzed (Participants) | 22 | 18 | 10 | 17 | 34 | 36
ug/mL | 54.8 (51.0) | 56.6 (34.0) | 81.4 (41.0) | 63.9 (30.0) | 106.0 (46.0) | 57.8 (31.0)

2. Primary Outcome: Time Taken to Reach Cmax (Tmax) - Parts A, B, D, and E
Description: Tmax is the time taken to reach the maximum observed serum nivolumab concentration (Cmax). Collected for Arm A, B, and D on Cycle 1 Day 1, Cycle 1 Day 2, Cycle 1 Day 4, Cycle 1 Day 8, Cycle 1 Day 15, and Cycle 1 Day 21. Collected for Arm E on Cycle 1 Day 1, Cycle 1 Day 2, Cycle 1 Day 4, Cycle 1 Day 8, Cycle 1 Day 15.
Time Frame: From first dose until approximately 21 days post first dose.
Population: as for outcome 1
Measure: Median (Full Range); unit: hours
Arm/Group | Part A - Group 1: Nivolumab + rHuPH20 SC 720mg | Part B - Group 2: Nivolumab SC 720mg | Part B - Group 3: Nivolumab + rHuPH20 SC 960mg | Part B - Group 4: Nivolumab SC 960mg | Part D: Nivolumab SC + rHuPH20 SC 1200mg Q4W | Part E: Nivolumab SC Co-Formulated With rHuPH20 600mg Q2W
Number analyzed (Participants) | 22 | 18 | 10 | 17 | 34 | 36
hours | 167 [47.0 to 357.0] | 167 [50.1 to 339.0] | 141 [47.2 to 333.0] | 168 [139.0 to 355.0] | 130 [44.5 to 317.0] | 130 [45.2 to 337.0]

3. Primary Outcome: Area Under the Time-Serum Nivolumab Concentration Curve (AUC (TAU)) - Parts A, B, D, and E
Description: AUC (TAU) is the area measured under the concentration-time curve taken over the dosing interval. Collected for Arm A, B, and D on Cycle 1 Day 1, Cycle 1 Day 2, Cycle 1 Day 4, Cycle 1 Day 8, Cycle 1 Day 15, and Cycle 1 Day 21. Collected for Arm E on Cycle 1 Day 1, Cycle 1 Day 2, Cycle 1 Day 4, Cycle 1 Day 8, Cycle 1 Day 15.
Time Frame: From first dose until approximately 21 days post first dose.
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ug/mL
Arm/Group | Part A - Group 1: Nivolumab + rHuPH20 SC 720mg | Part B - Group 2: Nivolumab SC 720mg | Part B - Group 3: Nivolumab + rHuPH20 SC 960mg | Part B - Group 4: Nivolumab SC 960mg | Part D: Nivolumab SC + rHuPH20 SC 1200mg Q4W | Part E: Nivolumab SC Co-Formulated With rHuPH20 600mg Q2W
Number analyzed (Participants) | 20 | 16 | 10 | 13 | 33 | 35
h*ug/mL | 24908 (53) | 27909 (36) | 40264 (45) | 32702 (31) | 53561 (40) | 15857 (30)

4. Primary Outcome: Observed Serum Nivolumab Concentration at the End of Dosing (Ctau) - Parts A, B, D, and E
Description: Ctau is the observed serum nivolumab concentration at the end of the dosing interval. Collected for Arma A, B, and D.
Time Frame: At the end of dosing interval of Cycle 1 - first dose (Day 21 for Parts A, B and D; Day 15 for Part E)
Population: All treated participants with available cycle 1 PK results in Parts A, B, D, and E. Pre-specified for data to be collected only in Parts A, B, D, and E.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Part A - Group 1: Nivolumab + rHuPH20 SC 720mg | Part B - Group 2: Nivolumab SC 720mg | Part B - Group 3: Nivolumab + rHuPH20 SC 960mg | Part B - Group 4: Nivolumab SC 960mg | Part D: Nivolumab SC + rHuPH20 SC 1200mg Q4W | Part E: Nivolumab SC Co-Formulated With rHuPH20 600mg Q2W
Number analyzed (Participants) | 20 | 16 | 10 | 13 | 33 | 35
ug/mL | 22.2 (86) | 26.9 (65) | 39.2 (67) | 34.8 (41) | 54.4 (49) | 43.6 (36)

5. Primary Outcome: Lowest Observed Serum Nivolumab Concentration (Ctrough) During Part C - Part A and B Crossover Participants to Part C
Description: Ctrough assessed during Part C. Ctrough is the lowest observed serum nivolumab concentration.
Time Frame: On Day 1 of Cycles 2, 3, 5, 9, 13, and 19 of Part C (Day 1 of Part C: up to 14 months from Baseline; each cycle was 28 days)
Population: All participants in Part C (who crossed over from Part A or B) with available PK results for each visit. Pre-specified for data to be reported for Part C crossover participants only. Participants are presented under their original treatment assignment.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Part A - Group 1: Nivolumab + rHuPH20 SC 720mg | Part B - Group 2: Nivolumab SC 720mg | Part B - Group 3: Nivolumab + rHuPH20 SC 960mg | Part B - Group 4: Nivolumab SC 960mg
Number analyzed (Participants) | 7 | 6 | 2 | 8
ug/mL
  Cycle 2 Day 1 | 115 (58) | 106 (42) | 124 (38) | 85.7 (48)
  Cycle 3 Day 1: number analyzed (Participants) | 7 | 5 | 2 | 3
  Cycle 3 Day 1 | 119 (51) | 118 (34) | 149 (42) | 104 (44)
  Cycle 5 Day 1: number analyzed (Participants) | 6 | 4 | 2 | 2
  Cycle 5 Day 1 | 149 (55) | 144 (66) | 192 (16) | 171 (8)
  Cycle 9 Day 1: number analyzed (Participants) | 6 | 2 | 1 | 2
  Cycle 9 Day 1 | 170 (55) | 138 (81) | 228 (NA) — Insufficient number of participants to calculate Geometric Coefficient of Variation. | 208 (38)
  Cycle 13 Day 1: number analyzed (Participants) | 4 | 3 | 1 | 2
  Cycle 13 Day 1 | 183 (34) | 113 (48) | 246 (NA) — Insufficient number of participants to calculate Geometric Coefficient of Variation. | 217 (16)
  Cycle 19 Day 1: number analyzed (Participants) | 0 | 1 | 0 | 1
  Cycle 19 Day 1 |  | 74.7 (NA) — Insufficient number of participants to calculate Geometric Coefficient of Variation. |  | 212 (NA) — Insufficient number of participants to calculate Geometric Coefficient of Variation.

6. Secondary Outcome: Number of Participants Experiencing Adverse Events (AEs)
Description: An Adverse Event (AE) is defined as any new untoward medical occurrence or worsening of a preexisting medical condition in a clinical investigation participant administered study treatment and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (such as an abnormal laboratory finding), symptom, or disease temporally associated with the use of study treatment, whether or not considered related to the study treatment.
Time Frame: From first dose until 100 days post last dose (up to approximately 70 months).
Population: All treated participants who received nivolumab subcutaneously (SC) and/or nivolumab intravenously (IV).
Measure: Count of Participants; unit: Participants
Groups:
- Part C - Nivolumab + rHuPH20 SC 1200mg Q4W (Crossover Participants From Parts A and B): Participants in Part A and Part B crossed over from nivolumab (BMS-936558) IV dosing (four [4] weeks after last IV dose) to nivolumab (BMS-986298) 1200 mg administered subcutaneously (SC) with recombinant human hyaluronidase (rHuPH20) manually by syringe every 4 weeks. Treatment continued until until Response Evaluation Criteria in Solid Tumors (RECIST) v.1.1 progression, unacceptable toxicity, withdrawal of consent, or completion of 104 weeks of treatment, whichever occured first.
Arm/Group | Part A - Group 1: Nivolumab + rHuPH20 SC 720mg | Part B - Group 2: Nivolumab SC 720mg | Part B - Group 3: Nivolumab + rHuPH20 SC 960mg | Part B - Group 4: Nivolumab SC 960mg | Part C - Nivolumab + rHuPH20 SC 1200mg Q4W (Crossover Participants From Parts A and B) | Part D: Nivolumab SC + rHuPH20 SC 1200mg Q4W | Part E: Nivolumab SC Co-Formulated With rHuPH20 600mg Q2W
Number analyzed (Participants) | 22 | 18 | 10 | 17 | 28 | 36 | 36
Participants | 22 | 18 | 10 | 17 | 27 | 36 | 36

7. Secondary Outcome: Number of Participants Experiencing Treatment Related Adverse Events (TRAEs)
Description: An Adverse Event (AE) is defined as any new untoward medical occurrence or worsening of a preexisting medical condition in a clinical investigation participant administered study treatment and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (such as an abnormal laboratory finding), symptom, or disease temporally associated with the use of study treatment, whether or not considered related to the study treatment. TRAEs are AEs where a reasonable causal relationship exists between study treatment administration and the AE.
Time Frame: From first dose until 100 days post last dose (up to approximately 70 months).
Population: All treated participants who received nivolumab subcutaneously (SC) and/or nivolumab intravenously (IV).
Measure: Count of Participants; unit: Participants
Arm/Group | Part A - Group 1: Nivolumab + rHuPH20 SC 720mg | Part B - Group 2: Nivolumab SC 720mg | Part B - Group 3: Nivolumab + rHuPH20 SC 960mg | Part B - Group 4: Nivolumab SC 960mg | Part C - Nivolumab + rHuPH20 SC 1200mg Q4W (Crossover Participants From Parts A and B) | Part D: Nivolumab SC + rHuPH20 SC 1200mg Q4W | Part E: Nivolumab SC Co-Formulated With rHuPH20 600mg Q2W
Number analyzed (Participants) | 22 | 18 | 10 | 17 | 28 | 36 | 36
Participants | 14 | 10 | 8 | 11 | 16 | 27 | 28

8. Secondary Outcome: Number of Participants Experiencing Serious Adverse Events (SAEs)
Description: A Serious Adverse Event (SAE) is defined as any untoward medical occurrence that, at any dose: (a) results in death, (b) is life-threatening (defined as an event in which the participant was at risk of death at the time of the event; it does not refer to an event which hypothetically might have caused death if it were more severe), and/ or (c) requires inpatient hospitalization or causes prolongation of existing hospitalization.
Time Frame: From first dose until 100 days post last dose (up to approximately 70 months).
Population: All treated participants who received nivolumab subcutaneously (SC) and/or nivolumab intravenously (IV).
Measure: Count of Participants; unit: Participants
Arm/Group | Part A - Group 1: Nivolumab + rHuPH20 SC 720mg | Part B - Group 2: Nivolumab SC 720mg | Part B - Group 3: Nivolumab + rHuPH20 SC 960mg | Part B - Group 4: Nivolumab SC 960mg | Part C - Nivolumab + rHuPH20 SC 1200mg Q4W (Crossover Participants From Parts A and B) | Part D: Nivolumab SC + rHuPH20 SC 1200mg Q4W | Part E: Nivolumab SC Co-Formulated With rHuPH20 600mg Q2W
Number analyzed (Participants) | 22 | 18 | 10 | 17 | 28 | 36 | 36
Participants | 12 | 10 | 4 | 11 | 11 | 19 | 25

9. Secondary Outcome: Number of Participants Experiencing Treatment Related Serious Adverse Events (TRSAEs)
Description: A Serious Adverse Event (SAE) is defined as any untoward medical occurrence that, at any dose: (a) results in death, (b) is life-threatening (defined as an event in which the participant was at risk of death at the time of the event; it does not refer to an event which hypothetically might have caused death if it were more severe), and/ or (c) requires inpatient hospitalization or causes prolongation of existing hospitalization. TRSAEs are SAEs where a reasonable causal relationship exists between study treatment administration and the SAE.
Time Frame: From first dose until 100 days post last dose (up to approximately 70 months).
Population: All treated participants who received nivolumab subcutaneously (SC) and/or nivolumab intravenously (IV).
Measure: Count of Participants; unit: Participants
Arm/Group | Part A - Group 1: Nivolumab + rHuPH20 SC 720mg | Part B - Group 2: Nivolumab SC 720mg | Part B - Group 3: Nivolumab + rHuPH20 SC 960mg | Part B - Group 4: Nivolumab SC 960mg | Part C - Nivolumab + rHuPH20 SC 1200mg Q4W (Crossover Participants From Parts A and B) | Part D: Nivolumab SC + rHuPH20 SC 1200mg Q4W | Part E: Nivolumab SC Co-Formulated With rHuPH20 600mg Q2W
Number analyzed (Participants) | 22 | 18 | 10 | 17 | 28 | 36 | 36
Participants | 1 | 1 | 0 | 2 | 0 | 3 | 1

10. Secondary Outcome: Number of Participants Experiencing Treatment Related Adverse Events (TRAEs) Leading to Discontinuation
Description: as for outcome 7
Time Frame: From first dose until 100 days post last dose (up to approximately 70 months).
Population: All treated participants who received nivolumab subcutaneously (SC) and/or nivolumab intravenously (IV).
Measure: Count of Participants; unit: Participants
Arm/Group | Part A - Group 1: Nivolumab + rHuPH20 SC 720mg | Part B - Group 2: Nivolumab SC 720mg | Part B - Group 3: Nivolumab + rHuPH20 SC 960mg | Part B - Group 4: Nivolumab SC 960mg | Part C - Nivolumab + rHuPH20 SC 1200mg Q4W (Crossover Participants From Parts A and B) | Part D: Nivolumab SC + rHuPH20 SC 1200mg Q4W | Part E: Nivolumab SC Co-Formulated With rHuPH20 600mg Q2W
Number analyzed (Participants) | 22 | 18 | 10 | 17 | 28 | 36 | 36
Participants | 2 | 1 | 1 | 2 | 0 | 4 | 2

11. Secondary Outcome: Number of Participants Who Died
Description: Number of participants who died due to any cause.
Time Frame: From randomization until data cutoff (up to approximately 70 months).
Population: All treated participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A - Group 1: Nivolumab + rHuPH20 SC 720mg | Part B - Group 2: Nivolumab SC 720mg | Part B - Group 3: Nivolumab + rHuPH20 SC 960mg | Part B - Group 4: Nivolumab SC 960mg | Part C - Nivolumab + rHuPH20 SC 1200mg Q4W (Crossover Participants From Parts A and B) | Part D: Nivolumab SC + rHuPH20 SC 1200mg Q4W | Part E: Nivolumab SC Co-Formulated With rHuPH20 600mg Q2W
Number analyzed (Participants) | 22 | 18 | 10 | 17 | 28 | 36 | 36
Participants | 18 | 14 | 8 | 14 | 17 | 25 | 30

12. Secondary Outcome: Number of Participants With Select Laboratory Changes From Baseline
Description: Laboratory parameters including hematology, chemistry, liver function, and renal function summarized using worst grade NCI CTCAE v.5 criteria. Baseline refers to evaluations with a date on or prior to the day of first dose of study treatment.
Time Frame: From first dose until 30 days post last dose (up to approximately 67 months and 20 days).
Population: All treated participants with baseline and at least one on treatment laboratory measurement.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A - Group 1: Nivolumab + rHuPH20 SC 720mg | Part B - Group 2: Nivolumab SC 720mg | Part B - Group 3: Nivolumab + rHuPH20 SC 960mg | Part B - Group 4: Nivolumab SC 960mg | Part C - Nivolumab + rHuPH20 SC 1200mg Q4W (Crossover Participants From Parts A and B) | Part D: Nivolumab SC + rHuPH20 SC 1200mg Q4W | Part E: Nivolumab SC Co-Formulated With rHuPH20 600mg Q2W
Number analyzed (Participants) | 21 | 16 | 10 | 16 | 28 | 36 | 36
Participants
  HEMOGLOBIN (g/L) | 13 | 7 | 3 | 8 | 15 | 12 | 12
  PLATELET COUNT (10^9/L) | 2 | 5 | 0 | 2 | 5 | 6 | 4
  LEUKOCYTES, LOCAL LAB (10^9/L) | 1 | 5 | 1 | 1 | 7 | 3 | 3
  ABSOLUTE NEUTROPHIL COUNT DRV. (10^9/L) | 2 | 2 | 1 | 2 | 5 | 2 | 3
  LYMPHOCYTES (ABSOLUTE) (10^9/L): number analyzed (Participants) | 0 | 3 | 0 | 4 | 5 | 4 | 3
  LYMPHOCYTES (ABSOLUTE) (10^9/L) |  | 3 |  | 2 | 2 | 2 | 3
  LYMPHOCYTES (ABSOLUTE), LOCAL LAB (10^9/L): number analyzed (Participants) | 21 | 13 | 10 | 11 | 28 | 32 | 33
  LYMPHOCYTES (ABSOLUTE), LOCAL LAB (10^9/L) | 10 | 9 | 5 | 5 | 12 | 7 | 16
  CREATININE, LOCAL LAB (umol/L) | 7 | 1 | 3 | 2 | 8 | 8 | 12
  ALKALINE PHOSPHATASE (ALP) LOCAL LAB (U/L): number analyzed (Participants) | 20 | 16 | 10 | 16 | 28 | 36 | 36
  ALKALINE PHOSPHATASE (ALP) LOCAL LAB (U/L) | 7 | 6 | 3 | 9 | 8 | 18 | 20
  ALANINE AMINOTRANSFERASE (ALT), LOCAL LAB (U/L) | 6 | 8 | 3 | 7 | 9 | 7 | 11
  ASPARTATE AMINOTRANSFERASE (AST), LOCAL LAB (U/L) | 5 | 9 | 4 | 6 | 6 | 11 | 14
  BILIRUBIN, TOTAL, LOCAL LAB (umol/L) | 2 | 6 | 1 | 2 | 5 | 4 | 6
  HYPERCALCEMIA (mmol/L): number analyzed (Participants) | 20 | 16 | 10 | 15 | 28 | 33 | 36
  HYPERCALCEMIA (mmol/L) | 1 | 1 | 1 | 2 | 2 | 6 | 3
  HYPERKALEMIA (mmol/L): number analyzed (Participants) | 21 | 16 | 10 | 15 | 28 | 36 | 36
  HYPERKALEMIA (mmol/L) | 7 | 4 | 4 | 2 | 9 | 7 | 9
  HYPERMAGNESEMIA (mmol/L): number analyzed (Participants) | 20 | 16 | 10 | 15 | 28 | 36 | 7
  HYPERMAGNESEMIA (mmol/L) | 0 | 0 | 0 | 0 | 0 | 0 | 0
  HYPERNATREMIA (mmol/L): number analyzed (Participants) | 21 | 16 | 10 | 15 | 28 | 36 | 36
  HYPERNATREMIA (mmol/L) | 2 | 1 | 1 | 2 | 5 | 4 | 3
  HYPOCALCEMIA (mmol/L): number analyzed (Participants) | 20 | 16 | 10 | 15 | 28 | 33 | 36
  HYPOCALCEMIA (mmol/L) | 5 | 2 | 2 | 2 | 2 | 4 | 5
  HYPOKALEMIA (mmol/L): number analyzed (Participants) | 21 | 16 | 10 | 15 | 28 | 36 | 36
  HYPOKALEMIA (mmol/L) | 1 | 1 | 1 | 1 | 3 | 3 | 5
  HYPOMAGNESEMIA (mmol/L): number analyzed (Participants) | 20 | 16 | 10 | 15 | 28 | 36 | 8
  HYPOMAGNESEMIA (mmol/L) | 5 | 1 | 1 | 3 | 3 | 2 | 2
  HYPONATREMIA (mmol/L): number analyzed (Participants) | 21 | 16 | 10 | 15 | 28 | 36 | 36
  HYPONATREMIA (mmol/L) | 8 | 4 | 5 | 3 | 9 | 9 | 13
  HYPOGLYCEMIA (mmol/L): number analyzed (Participants) | 20 | 16 | 10 | 16 | 28 | 34 | 35
  HYPOGLYCEMIA (mmol/L) | 1 | 1 | 0 | 1 | 2 | 2 | 1
  ALBUMIN, LOCAL LAB (g/L): number analyzed (Participants) | 20 | 16 | 10 | 16 | 0 | 36 | 9
  ALBUMIN, LOCAL LAB (g/L) | 6 | 6 | 3 | 2 |  | 13 | 5
  ACTIVATED PARTIAL THROMBOPLASTIN TIME (sec): number analyzed (Participants) | 3 | 8 | 0 | 8 | 0 | 4 | 8
  ACTIVATED PARTIAL THROMBOPLASTIN TIME (sec) | 1 | 2 |  | 1 |  | 2 | 1
  FIBRINOGEN (g/L): number analyzed (Participants) | 2 | 9 | 0 | 8 | 0 | 6 | 11
  FIBRINOGEN (g/L) | 0 | 0 |  | 0 |  | 0 | 0

13. Secondary Outcome: Number of Participants Experiencing Any Select Adverse Events Within the Hypersensitivity/Infusion Reaction Category and Broad Standardized MedDRA Query (SMQ) of Anaphylactic Reaction Occurring Within 2 Days of Study Drug Administration
Description: as for outcome 6
Time Frame: From first dose until 2 days post last dose (up to approximately 66 months and 22 days).
Population: All treated participants who received nivolumab subcutaneously (SC) and/or nivolumab intravenously (IV).
Measure: Count of Participants; unit: Participants
Arm/Group | Part A - Group 1: Nivolumab + rHuPH20 SC 720mg | Part B - Group 2: Nivolumab SC 720mg | Part B - Group 3: Nivolumab + rHuPH20 SC 960mg | Part B - Group 4: Nivolumab SC 960mg | Part C - Nivolumab + rHuPH20 SC 1200mg Q4W (Crossover Participants From Parts A and B) | Part D: Nivolumab SC + rHuPH20 SC 1200mg Q4W | Part E: Nivolumab SC Co-Formulated With rHuPH20 600mg Q2W
Number analyzed (Participants) | 22 | 18 | 10 | 17 | 28 | 36 | 36
Participants
  Nivolumab administered subcutaneously (SC) +/- rHuPH20 | 1 | 1 | 0 | 0 | 4 | 3 | 8
  Nivolumab administered intravenously (IV): number analyzed (Participants) | 19 | 16 | 10 | 14 | 0 | 0 | 0
  Nivolumab administered intravenously (IV) | 2 | 2 | 1 | 2 |  |  |

14. Secondary Outcome: Number of Participants With Anti-Nivolumab Antibodies (ADAs) and Neutralizing Antibodies
Description: Anti-drug antibody (ADA) Positive: A participant with at least one ADA-positive sample relative to baseline (ADA negative at baseline or ADA titer to be at least 4-fold or greater (>=) than baseline positive titer) at any time after initiation of treatment; Neutralizing Positive: At least one ADA-positive sample with neutralizing antibodies detected post-baseline.
  Baseline ADA Positive: A participant with a baseline ADA-positive sample. Baseline refers to evaluations with a date on or prior to the day of first dose of study treatment.
Time Frame: At baseline and up to 100 days post last dose (up to approximately 70 months).
Population: Immunogenicity Evaluable Participants: All treated participants in Parts A-E who have a baseline and at least 1 post-baseline immunogenicity assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A - Group 1: Nivolumab + rHuPH20 SC 720mg | Part B - Group 2: Nivolumab SC 720mg | Part B - Group 3: Nivolumab + rHuPH20 SC 960mg | Part B - Group 4: Nivolumab SC 960mg | Part C - Nivolumab + rHuPH20 SC 1200mg Q4W (Crossover Participants From Parts A and B) | Part D: Nivolumab SC + rHuPH20 SC 1200mg Q4W | Part E: Nivolumab SC Co-Formulated With rHuPH20 600mg Q2W
Number analyzed (Participants) | 21 | 18 | 10 | 17 | 28 | 36 | 35
Participants
  ANTI-DRUG ANTIBODY (ADA) POSITIVE | 7 | 5 | 3 | 0 | 7 | 5 | 10
  NEUTRALIZING POSITIVE | 0 | 0 | 0 | 0 | 0 | 0 | 0
  BASELINE ANTI-DRUG ANTIBODY (ADA) POSITIVE | 2 | 0 | 2 | 0 | 2 | 1 | 1

ADVERSE EVENTS:
Time Frame: All-cause Mortality was collected from randomization until the data cutoff date (approximately 70 months). SAEs and Other AEs were collected from the first dose until 100 days post the last dose (up to approximately 70 months).
Description: All-Cause Mortality, SAEs and Other AEs refer to all the participants who were treated with study medicine. For Cohort C crossover participants, data were reported according to the group from which they crossed over as prespecified.
Groups:
- PART A - GRP 1 CROSSOVER to PART C: Some participants in Part A crossed over to Part C, four weeks after their last nivolumab IV dose to receive nivolumab (BMS-986298) 1200 mg administered subcutaneously (SC) with recombinant human hyaluronidase (rHuPH20) manually by syringe every 4 weeks. Treatment continued until Response Evaluation Criteria in Solid Tumors (RECIST) v.1.1 progression, unacceptable toxicity, withdrawal of consent, or completion of 104 weeks of treatment, whichever occured first.
- PART B - GRP 2 CROSSOVER to PART C: Some participants in Part B - Group 2 crossed over to Part C, four weeks after their last nivolumab IV dose to receive nivolumab (BMS-986298) 1200 mg administered subcutaneously (SC) with recombinant human hyaluronidase (rHuPH20) manually by syringe every 4 weeks. Treatment continued until Response Evaluation Criteria in Solid Tumors (RECIST) v.1.1 progression, unacceptable toxicity, withdrawal of consent, or completion of 104 weeks of treatment, whichever occured first.
- PART B - GRP 3 CROSSOVER to PART C: Some participants in Part B - Group 3 crossed over to Part C, four weeks after their last nivolumab IV dose to receive nivolumab (BMS-986298) 1200 mg administered subcutaneously (SC) with recombinant human hyaluronidase (rHuPH20) manually by syringe every 4 weeks. Treatment continued until Response Evaluation Criteria in Solid Tumors (RECIST) v.1.1 progression, unacceptable toxicity, withdrawal of consent, or completion of 104 weeks of treatment, whichever occured first.
- PART B - GRP 4 CROSSOVER to PART C: Some participants in Part B - Group 4 crossed over to Part C, four weeks after their last nivolumab IV dose to receive nivolumab (BMS-986298) 1200 mg administered subcutaneously (SC) with recombinant human hyaluronidase (rHuPH20) manually by syringe every 4 weeks. Treatment continued until Response Evaluation Criteria in Solid Tumors (RECIST) v.1.1 progression, unacceptable toxicity, withdrawal of consent, or completion of 104 weeks of treatment, whichever occured first.
Arm/Group | Part A - Group 1: Nivolumab + rHuPH20 SC 720mg | PART A - GRP 1 CROSSOVER to PART C | Part B - Group 2: Nivolumab SC 720mg | PART B - GRP 2 CROSSOVER to PART C | Part B - Group 3: Nivolumab + rHuPH20 SC 960mg | PART B - GRP 3 CROSSOVER to PART C | Part B - Group 4: Nivolumab SC 960mg | PART B - GRP 4 CROSSOVER to PART C | Part D: Nivolumab SC + rHuPH20 SC 1200mg Q4W | Part E: Nivolumab SC Co-Formulated With rHuPH20 600mg Q2W
All-Cause Mortality (participants affected / at risk) | 18/22 | 6/9 | 14/18 | 2/6 | 8/10 | 4/5 | 14/17 | 5/8 | 25/36 | 30/36
Serious Adverse Events (participants affected / at risk) | 12/22 | 4/9 | 10/18 | 1/6 | 4/10 | 2/5 | 11/17 | 4/8 | 19/36 | 25/36
Other Adverse Events (participants affected / at risk) | 22/22 | 9/9 | 18/18 | 6/6 | 10/10 | 5/5 | 17/17 | 8/8 | 34/36 | 35/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A - Group 1: Nivolumab + rHuPH20 SC 720mg (N=22) | PART A - GRP 1 CROSSOVER to PART C (N=9) | Part B - Group 2: Nivolumab SC 720mg (N=18) | PART B - GRP 2 CROSSOVER to PART C (N=6) | Part B - Group 3: Nivolumab + rHuPH20 SC 960mg (N=10) | PART B - GRP 3 CROSSOVER to PART C (N=5) | Part B - Group 4: Nivolumab SC 960mg (N=17) | PART B - GRP 4 CROSSOVER to PART C (N=8) | Part D: Nivolumab SC + rHuPH20 SC 1200mg Q4W (N=36) | Part E: Nivolumab SC Co-Formulated With rHuPH20 600mg Q2W (N=36)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2
Atrial flutter (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrial thrombosis (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Myocarditis (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Intestinal perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Subileus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Death (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
General physical health deterioration (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Cholangitis (Hepatobiliary disorders) | 0 | 0 | 2 | 1 | 0 | 0 | 1 | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hepatitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Contrast media allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3
COVID-19 pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Empyema (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Escherichia infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Lung abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 2 | 2 | 3 | 2 | 0 | 2
Pseudomonal sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Lipase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Infected metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 1 | 5 | 0 | 0 | 0 | 4 | 1 | 4 | 7
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tumour fistulisation (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tumour obstruction (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Brain stem haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cerebellar haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Epilepsy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Ischaemic cerebral infarction (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Spinal cord compression (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Device dislocation (Product Issues) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tubulointerstitial nephritis (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pemphigoid (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Part A - Group 1: Nivolumab + rHuPH20 SC 720mg (N=22) | PART A - GRP 1 CROSSOVER to PART C (N=9) | Part B - Group 2: Nivolumab SC 720mg (N=18) | PART B - GRP 2 CROSSOVER to PART C (N=6) | Part B - Group 3: Nivolumab + rHuPH20 SC 960mg (N=10) | PART B - GRP 3 CROSSOVER to PART C (N=5) | Part B - Group 4: Nivolumab SC 960mg (N=17) | PART B - GRP 4 CROSSOVER to PART C (N=8) | Part D: Nivolumab SC + rHuPH20 SC 1200mg Q4W (N=36) | Part E: Nivolumab SC Co-Formulated With rHuPH20 600mg Q2W (N=36)
Anaemia (Blood and lymphatic system disorders) | 5 | 1 | 6 | 1 | 3 | 2 | 2 | 1 | 3 | 7
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Ear discomfort (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 3
Hyperthyroidism (Endocrine disorders) | 3 | 2 | 0 | 0 | 0 | 0 | 3 | 1 | 6 | 1
Hypothyroidism (Endocrine disorders) | 2 | 2 | 2 | 2 | 0 | 0 | 1 | 1 | 8 | 8
Eye pruritus (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Lacrimation increased (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 3 | 1 | 2 | 1 | 0 | 0 | 3 | 0 | 3 | 5
Abdominal pain upper (Gastrointestinal disorders) | 3 | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 1 | 6
Autoimmune colitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chronic gastritis (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 2 | 2 | 3 | 0 | 2 | 0 | 1 | 0 | 5 | 5
Diarrhoea (Gastrointestinal disorders) | 5 | 2 | 4 | 3 | 1 | 1 | 4 | 2 | 4 | 6
Dry mouth (Gastrointestinal disorders) | 1 | 1 | 3 | 2 | 0 | 0 | 1 | 0 | 0 | 4
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 5 | 1 | 3 | 1 | 2 | 1 | 3 | 2 | 2 | 8
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 1 | 2
Subileus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 4 | 1 | 2 | 2 | 0 | 0 | 3 | 1 | 3 | 2
Asthenia (General disorders) | 5 | 2 | 7 | 2 | 0 | 0 | 2 | 1 | 2 | 8
Chest pain (General disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Chills (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Facial pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 5 | 3 | 3 | 2 | 1 | 1 | 3 | 2 | 6 | 6
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Injection site erythema (General disorders) | 4 | 2 | 1 | 1 | 6 | 4 | 2 | 2 | 6 | 1
Injection site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Injection site pruritus (General disorders) | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 1 | 0
Injection site reaction (General disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 10
Injection site swelling (General disorders) | 3 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nodule (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Oedema peripheral (General disorders) | 7 | 3 | 2 | 1 | 2 | 1 | 0 | 0 | 3 | 1
Pain (General disorders) | 1 | 1 | 0 | 0 | 1 | 1 | 1 | 1 | 2 | 0
Pyrexia (General disorders) | 5 | 2 | 6 | 1 | 0 | 0 | 0 | 0 | 3 | 3
Secretion discharge (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Cholestasis (Hepatobiliary disorders) | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic cytolysis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Hypertransaminasaemia (Hepatobiliary disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4
Candida infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Ear infection (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0
Hordeolum (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 2 | 2 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 2
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Norovirus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Oral candidiasis (Infections and infestations) | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 3
Pilonidal disease (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 1 | 1
Rash pustular (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Skin infection (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 3 | 3
Urinary tract infection (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 3
Vulvovaginal candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0
Immunisation reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Injection related reaction (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 4 | 5
Amylase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 1 | 2 | 1 | 1 | 0 | 1 | 0 | 3 | 6
Blood albumin decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 0 | 4 | 1 | 0 | 0 | 0 | 0 | 1 | 3
Blood bilirubin increased (Investigations) | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 1 | 1
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 6
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 0 | 2 | 1 | 0 | 0 | 1 | 0 | 2 | 2
Hepatic enzyme increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lipase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0
Protein total decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 3 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Weight increased (Investigations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 3 | 3
Hyperamylasaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Hyperlipasaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Underweight (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 4 | 2 | 2 | 0 | 0 | 5 | 2 | 5 | 10
Arthritis (Musculoskeletal and connective tissue disorders) | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 1 | 0 | 0 | 1 | 1 | 3 | 3 | 5 | 5
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ligament pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 1 | 1 | 2 | 1 | 1 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 2 | 1 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 1
Rib deformity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 2 | 0
Dizziness (Nervous system disorders) | 2 | 2 | 0 | 0 | 1 | 1 | 2 | 1 | 2 | 0
Dizziness postural (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 1
Headache (Nervous system disorders) | 3 | 2 | 0 | 0 | 0 | 0 | 4 | 2 | 2 | 0
Monoparesis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1
Neuropathy peripheral (Nervous system disorders) | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1
Agitation (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Depressed mood (Psychiatric disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Insomnia (Psychiatric disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Haematuria (Renal and urinary disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Micturition urgency (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Asthma late onset (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 1 | 0 | 0 | 0 | 4 | 3 | 3 | 4
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 2 | 0 | 0 | 0 | 4 | 2 | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 1 | 1 | 1 | 0 | 3 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Lividity (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nail dystrophy (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 2 | 2 | 1 | 1 | 0 | 1 | 1 | 8 | 9
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 2 | 1 | 1 | 0 | 2 | 2 | 4 | 4
Rash erythematous (Skin and subcutaneous tissue disorders) | 3 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 1 | 2
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 1 | 1 | 1 | 1 | 1 | 0 | 1 | 1 | 1 | 1
Granulomatous lymphadenitis (Blood and lymphatic system disorders) | 1/13 | 0 | 0/12 | 0 | 0/5 | 0 | 0/9 | 0 | 0 | 0
Lymph node pain (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac failure chronic (Cardiac disorders) | 1/13 | 0 | 0/12 | 0 | 0/5 | 0 | 0/9 | 0 | 0 | 0
Diplopia (Eye disorders) | 1/13 | 0 | 0/12 | 0 | 0/5 | 0 | 0/9 | 0 | 0 | 0
Dry eye (Eye disorders) | 1/13 | 0 | 0/12 | 0 | 0/5 | 0 | 0/9 | 0 | 0 | 0
Periorbital swelling (Eye disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gait disturbance (General disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site irritation (General disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Folliculitis (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tooth abscess (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood folate decreased (Investigations) | 1/13 | 0 | 0/12 | 0 | 0/5 | 0 | 0/9 | 0 | 0 | 0
Thyroxine free increased (Investigations) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fluid retention (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gout (Metabolism and nutrition disorders) | 1/13 | 0 | 0/12 | 0 | 0/5 | 0 | 0/9 | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Coccydynia (Musculoskeletal and connective tissue disorders) | 1/13 | 0 | 0/12 | 0 | 0/5 | 0 | 0/9 | 0 | 0 | 0
Hypercreatinaemia (Musculoskeletal and connective tissue disorders) | 1/13 | 0 | 0/12 | 0 | 0/5 | 0 | 0/9 | 0 | 0 | 0
Osteopenia (Musculoskeletal and connective tissue disorders) | 1/13 | 0 | 0/12 | 0 | 0/5 | 0 | 0/9 | 0 | 0 | 0
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 1/13 | 0 | 0/12 | 0 | 0/5 | 0 | 0/9 | 0 | 0 | 0
Burning sensation (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperaesthesia (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 1/13 | 0 | 0/12 | 0 | 0/5 | 0 | 0/9 | 0 | 0 | 1
Motor dysfunction (Nervous system disorders) | 1/13 | 0 | 0/12 | 0 | 0/5 | 0 | 0/9 | 0 | 0 | 0
Sciatica (Nervous system disorders) | 1/13 | 0 | 0/12 | 0 | 0/5 | 0 | 0/9 | 0 | 0 | 0
Tremor (Nervous system disorders) | 1/13 | 0 | 0/12 | 0 | 0/5 | 0 | 0/9 | 0 | 0 | 0
Device dislocation (Product Issues) | 1/13 | 0 | 0/12 | 0 | 0/5 | 0 | 0/9 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Delirium (Psychiatric disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sleep disorder (Psychiatric disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dysuria (Renal and urinary disorders) | 1/13 | 0 | 0/12 | 0 | 0/5 | 0 | 0/9 | 0 | 1 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1/13 | 0 | 0/12 | 0 | 0/5 | 0 | 0/9 | 0 | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1/13 | 0 | 0/12 | 0 | 0/5 | 0 | 0/9 | 0 | 0 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1/13 | 0 | 0/12 | 0 | 0/5 | 0 | 0/9 | 0 | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1/13 | 0 | 0/12 | 0 | 0/5 | 0 | 0/9 | 0 | 0 | 1
Skin disorder (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin mass (Skin and subcutaneous tissue disorders) | 1/13 | 0 | 0/12 | 0 | 0/5 | 0 | 0/9 | 0 | 0 | 0
Haemorrhage (Vascular disorders) | 1/13 | 0 | 0/12 | 0 | 0/5 | 0 | 0/9 | 0 | 0 | 0
Hypotension (Vascular disorders) | 1/13 | 0 | 0/12 | 0 | 0/5 | 0 | 0/9 | 0 | 0 | 0
Vena cava thrombosis (Vascular disorders) | 1/13 | 0 | 0/12 | 0 | 0/5 | 0 | 0/9 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-08): https://cdn.clinicaltrials.gov/large-docs/18/NCT03656718/Prot_SAP_000.pdf